CLINICAL TRIAL: NCT05339451
Title: Blood and Tissue Markers for Improving Diagnosis and Prognosis of Endometriosis. a Prospective Multicenter Nationwide Study. (ENDOBIO)
Brief Title: Blood and Tissue Markers for Improving Diagnosis and Prognosis of Endometriosis. (ENDOBIO)
Acronym: ENDOBIO
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other); Södersjukhuset (Stockholm South General Hospital) (Unknown); Akademiska University Hospital, Uppsala, Sweden (Unknown)
Responsible Party: Sponsor
Other Study IDs: K 2022-2797
Record Dates: First submitted 2022-04-05; First posted 2022-04-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
Keywords: endometriosis; biomarkers
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Severe/Deep infiltrating endometriosis: Endometriosis stage III/IV according to rASRM.
  Interventions: Diagnostic Test: Blood biomarkers
- Minimal/mild endometriosis: Endometriosis stage I/II according to rASRM
  Interventions: Diagnostic Test: Blood biomarkers
- Controls: Women operated for other benign gynecological diseases and have no signs of endometriosis perioperatively.
  Interventions: Diagnostic Test: Blood biomarkers

INTERVENTIONS:
Diagnostic Test: Blood biomarkers — Blood biomarkers in plasma and serum.

SUMMARY:
Endometriosis is a chronic, benign, estrogen-dependent disease characterized by endometrial tissue that is implanted outside the uterus into the ovaries, intestines, or peritoneum but also outside the pelvis. It is a common disease that affects 7-10% of women around the world. The most common symptoms are pain and infertility. The diagnosis is histological after removal of lesions with laparoscopy (sensitivity 94%, specificity 79%), and treatment is symptomatic.

At present, there is not a laboratory test that allows early and adequate diagnosis of endometriosis and therefore it can take up to 10 years for a patient to be diagnosed and patients often suffer from the disease.

The purpose of our study is to investigate biomarkers associated with endometriosis and prove their use in the diagnosis and staging of endometriosis. The biomarkers will be studied even in relationship to clinical manifestations of the disease, as markers of relapse and as fertility markers. Meanwhile, quality of life of patients with advanced stages of endometriosis postoperatively will be studied.

ELIGIBILITY:
IInclusion Criteria:

* women of reproductive age (18-45) who are operated because of suspected endometriosis (dysmenorrhea, dyspareunia, infertility, etc.) (patient group)
* women of reproductive age (18-45) who are operated for other benign gynecological causes with laparoscopy (ovarian cysts, sterilization, fibroids, etc.) and are found without macroscopic endometriosis perioperatively and confirmed with blind biopsies (control group
* talk swedish or english in order to complete questionnaires and give informed consent for their participation in the study.

Exclusion Criteria:

* BMI> 40
* postmenopausal women
* premature ovarian failure
* pelvic inflammatory disease (PID)
* current or previous malignancy
* pregnancy and 6 months postpartum
* corticosteroids in the last 3 months
* pituitary, kidney, liver, adrenal disease
* endometrial hyperplasia or endometrial polyp
* cardiovascular or systemic inflammatory diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited in several gynecological clinics around Sweden. A total of 345 women of reproductive age will be included in the study according to the power calculation. 115 patients who are operated on due to deep infiltrating endometriosis or rASRM III-IV in national endometriosis centers in Sweden, 115 patients who are diagnosed during surgery with early-stage endometriosis (rASRM I-II) and 115 patients who are controls, who are operated on for others benign gynecological diseases (fibroids, ovarian cysts, chronic abdominal pain, sterilization) and have no signs of endometriosis perioperatively.
Sampling Method: Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of blood biomarkers panel for the diagnosis of endometriosis with sensitivity 94% | Preoperative
  Blood biomarkers as endometriosis diagnostic tests
Change in blood biomarkers levels 3-6 months postoperative in patients with severe endometriosis. | 3-6 months postoperative in the severe/DIE group
  Blood biomarkers as a relapse marker
Measurement of blood biomarkers panel for the diagnosis of endometriosis with specificity 79% | Preoperative
  Blood biomarkers as endometriosis diagnostic tests

SECONDARY OUTCOMES:
Quality of life of patients undergoing surgery for DIE | Preoperative and 3-6 months postoperative in the severe/DIE group
  Endometriosis Health Profile 30 Questionnaire
Achieved pregnancy postoperative | One year postoperative
  Positive pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Kenny Rodriguez-Wallberg, Professor, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Karolinska Universitetssjukhus Huddinge, Stockholm, Huddinge
  - Södersjukhuset Kvinnokliniken, Stockholm, Stockholm County
  - Akademiska Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: No